CLINICAL TRIAL: NCT03306459
Title: Hospital Clínic Barcelona
Brief Title: Psychological Traits, Sexuality and Quality of Life in Patients With Polycystic Ovary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Camil Castelo-Branco, Professor, Hospital Clinic of Barcelona
Other Study IDs: B/2017/0614
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; Quality of life; Sexuality; Psychological traits
MeSH Terms: conditions — Polycystic Ovary Syndrome; Sexuality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/PCOS: The authors will select 30 PCOS patients who met the more strict and conservative Rotterdam diagnostic criteria (Rotterdam phenotype A) which include the presence of oligo-anovulation (cycles lasting >35 days or amenorrhea) and hyperandrogenemia /hyperandrogenism (hirsutism or obvious acne or pronounced alopecia). All patients should have bilateral polycystic ovaries morphology on ultrasound. Additionally, the authors have decided to enroll PCOS patients that are all without pregnancy desire at the moment they fill out the questionnaires, in order to control for the potential confounding role of infertility on psychological outcomes. Different pituitary, adrenal, ovarian, thyroid or metabolic diseases will be excluded
  Interventions: Diagnostic Test: SF-36 (Short Form Health Survey)
- 2/CONTROL: The authors will enroll a control group of 30 women, age- matched with the PCOS women, from consecutive women controlled in the same outpatient clinic who met the following inclusion criteria: history of irregular menstrual cycle in absence of severe gynecologic and non-gynecologic diseases. This PCOS sample will be entirely constituted by women with no pregnancy desire; therefore, with the aim to limit the potential effect of the unfulfilled wish to conceive in the final results; additionally, infertile women will not admitted into the control group.
  Interventions: Diagnostic Test: SF-36 (Short Form Health Survey)

INTERVENTIONS:
Diagnostic Test: SF-36 (Short Form Health Survey) — Symptom Checklist-90-Revision (SCL-90-R): self-report questionnaire of 90 items on a 5-point Likert scale clustered in 9 primary scales (somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation and psychoticism).
  State-Trait-Anger-Expression-Inventory, version 2 (STAXI-2): self-report questionnaire of 57-items on a 4-point scale distributed in different dimensions: State-Anger, Trait-Anger Expression Anger (in-out) and Anger Control (in-out) Short Form Health Survey (SF-36), an instrument composed by 8 subscales: Physical Functioning, Physical Role Function, Bodily Pain, General Health, Vitality, Social Functioning, Emotional Role Function and Mental Health.
  Female Sexual Function Index (FSFI) a 19-item self-report measure of female sexual function providing scores on 6 domains (desire, arousal, lubrication, orgasm, satisfaction, pain) as well as a total score.
  Other Names: Female Sexual Function Index; Symptom Checklist-90-R; State-Trait-Anger-Expression-Inventory

SUMMARY:
A prospective assessment of psychological characteristics, quality of life and sexuality in naïve patients.

DETAILED DESCRIPTION:
This project with PCOS patients include an assessment of quality of life and sexuality in naïve patients.

Hypothesizing that PCOS women would show higher rates of psychological alterations, this study is aimed to investigate the association between polycystic ovary syndrome (PCOS) and psychological disturbances, including anger and to analyze whether the biochemical/phenotypical features of PCOS may play a role in the type and severity of psychological disorders.

ELIGIBILITY:
Inclusion Criteria:

PCOS patients without gestational desire who met the following criteria

* Oligomenorrhea (cycles lasting >35 days) or amenorrhea (no periods in 6 months)
* Hyperandrogenemia/hyperandrogenism Hirsutism Ferriman-Gallwey score > 12 Obvious acne or pronounced alopecia Androgen levels over normal female range

Exclusion Criteria:

* Prior psychiatric diagnosis
* Current use of psychiatric medications
* Difficulties with language comprehension in case of non-nationals.
* Yatrogenic hirsutism,
* Other endocrine deseases with hyperandrogenism or that may influence the final results Ovarian or adrenal neoplasia Prolactinoma Cushing's syndrome Congenital adrenal hyperplasia Diabetes mellitus Thromboembolic disease
* Patients who had received any drug therapy for hirsutism over the last 6 months

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The authors will select 30 PCOS patients who met the more strict and conservative Rotterdam diagnostic criteria (Rotterdam phenotype A)
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01-09 (Estimated); Primary Completion 2019-01-09 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | january 9th 2018-january 9th 2019
  results of SF-36

SECONDARY OUTCOMES:
Sexuality | january 9th 2018-january 9th 2019
  Results of FSFI
Psychological distress | january 9th 2018-january 9th 2019
  Results of Symptom Checklist-90-Revision (SCL-90-R)
Anger and aggressiveness | january 9th 2018-january 9th 2019
  results of State-Trait-Anger-Expression-Inventory, version 2 (STAXI-2)

OTHER OUTCOMES:
Biochemical markers | january 9th 2018-january 9th 2019
  Results of blood tests including biochemistry and hormones analysis
Phenotipical traits | january 9th 2018-january 9th 2019
  Record of hirsutism, acne, alopecia, and other hyperandrogenic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Camil Castelo-Branco, MD PhD, Study Director — Hospital Clínic. University of Barcelona
Locations (1):
- Hospital Clínic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naumova I, Castelo-Branco C, Casals G. Psychological Issues and Sexual Function in Women with Different Infertility Causes: Focus on Polycystic Ovary Syndrome. Reprod Sci. 2021 Oct;28(10):2830-2838. doi: 10.1007/s43032-021-00546-x. Epub 2021 Mar 24. PMID 33763818